CLINICAL TRIAL: NCT05360563
Title: Effects of a Home-based Exercise Program on the Functional Sequelae of Patients With the Post-COVID-19 Condition: A Randomized Controlled Trial
Brief Title: Home-based Exercise Program in Patients With the Post-COVID-19 Condition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5.052.767
Record Dates: First submitted 2022-05-02; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Long COVID; Post-acute COVID-19 Syndrome
Keywords: Exercise; Telemedicine; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical training group (Experimental): In addition to receive regular medical care, the physical training group will participate in a tailored home-based exercise program (remotely supervised by healthcare professionals).
  Interventions: Other: Home-based physical training
- Control group (No Intervention): The control group will receive regular medical care.

INTERVENTIONS:
Other: Home-based physical training — Patients allocated to this group will participate in a 16-week home-based physical training program, structured in three weekly sessions of aerobic and muscle strengthening exercises (which also have components that stimulate flexibility and balance). A third of the weekly physical training sessions will be supervised via telemedicine (with video call) by a clinical exercise specialist, but all patients will have illustrated exercise booklets and a full-time remote support service available for the remaining sessions (via text or voice messages).
  Arms: Physical training group

SUMMARY:
The management of the sequelae of COVID-19 is described as the next great challenge of global public health. Multiple symptoms may compose the clinical picture of these patients (eg, fatigue, dyspnea, cognitive dysfunction, myalgia and others), persisting for more than a year and frequently causing clinically important functional impairment. Thus, a clinical trial will be conducted to investigate the effects of a remotely supervised home-based exercise program on functional sequelae of patients diagnosed with the post-COVID-19 condition (also known as Long COVID).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnostic history confirmed by real-time reverse transcription-polymerase chain reaction (RT-PCR) or rapid antigen test (with clinical presentations of moderate to critical severity).
* Diagnosis of post-COVID-19 condition according to World Health Organization criteria.
* Present ≥1 symptoms at study admission, including dyspnea, fatigue, muscle weakness and/or musculoskeletal pain.
* Have internet access at home.

Exclusion Criteria:

* Being under clinical or experimental treatment for the post-COVID-19 condition.
* Any physical disabilities that could hamper physical testing and exercise program.
* Patients with major neuropsychiatric disorders (eg, dementia or severe depression).
* Patients with chronic kidney disease who are in need of hemodialysis.
* Solid organ transplant patients.
* Complex ventricular arrhythmias, atrial fibrillation or complete heart block.
* Recent malignant neoplasm.
* Recent deep venous thromboembolism.
* Acute pulmonary embolism or pulmonary infarction.
* Uncontrolled hypertension.
* Uncontrolled type II diabetes.
* Uncontrolled vestibular disorders.
* Acute infections.
* Pregnancy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in functional fitness assessed by distance walked (m) in the six-minute walk test (6MWT) at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.

SECONDARY OUTCOMES:
Change from baseline in six-minute walk work (kg.km) assessed by 6MWT at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in maximal inspiratory muscle strength (cmH2O) assessed by POWERbreathe device at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in forced vital capacity (FVC; L) assessed on spirometry at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in forced expiratory volume in 1 second (FEV1; L) assessed on spirometry at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in FEV1/FVC ratio (%) assessed on spirometry at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in peak expiratory flow (L/s) assessed on spirometry at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in peak inspiratory flow (L/s) assessed on spirometry at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in muscle strength (kgf) assessed by handgrip test at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in muscle function (number of repetitions) assessed by the 1-minute sit-to-stand test (1'STST) at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in functional symptom burden (arb. unit) assessed by a weekly composite at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.
Change from baseline in functional capacity (from 0 to 4 degrees of functional limitation) assessed by the post-COVID-19 functional status (PCFS) scale at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.
Change from baseline in physical activity levels (min/week of MVPA) assessed by the international physical activity questionnaires (IPAQ) at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in fatigue levels (from 0 to 33 points) assessed by the Chalder fatigue scale (CFQ) at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.
Change from baseline in executive functions (z-score) assessed in a battery of cognitive tests at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in learning and memory (z-score) assessed in a battery of cognitive tests at 16 weeks. | At baseline and after 16 weeks
  Higher score means better outcome.
Change from baseline in total body weight (kg) at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.
Change from baseline in waist circumference (cm) at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.
Change from baseline in hip circumference (cm) at 16 weeks. | At baseline and after 16 weeks
  Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, Brazil